CLINICAL TRIAL: NCT01952522
Title: Comparison of Two Rehabilitation Programs to Improve Walking in Community-dwelling People After Stroke
Brief Title: Effects of a Walking Intervention With Additional Weights on the Unaffected Leg in People After Stroke
Acronym: ANANTA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Collaborators: Centre Hospitalier Sainte Anne, Paris (Unknown); Département d'Epidémiologie Clinique, Hôpital Hôtel-Dieu, Paris (Unknown); URC-CIC Paris Descartes Necker Cochin (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: P110702
Record Dates: First submitted 2013-05-03; First posted 2013-09-30 (Estimated); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Stroke; Hemiparesis
Keywords: Resistance training; Walking; Weight bearing
MeSH Terms: conditions — Stroke; Paresis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Weighted brace (Experimental)
  Interventions: Behavioral: Weighted brace
- non weighted brace (Placebo Comparator)
  Interventions: Behavioral: Non weighted brace

INTERVENTIONS:
Behavioral: Weighted brace — People will have to wear all the day additional weights (between 2 and 4 kilograms) at the nonparetic ankle during 3 months
  Arms: Weighted brace
Behavioral: Non weighted brace — People will be given a brace with no weight they will have to wear all the day during three months.
  Arms: non weighted brace

SUMMARY:
This study is designed to determine if adding daily weighted braces on the unaffected ankle may benefit to patient who have returned home compare to a placebo intervention (ankle brace without weight).

DETAILED DESCRIPTION:
Improve walking ability in people after stroke is a key objective for rehabilitation. Once the rehabilitation period is finished, a reduction of functional and motor abilities is often observed in subjects when they returned home.

This study will examine if loading daily the non paretic leg with additional weights will improve walking abilities. This study will enroll 100 people who had a stroke > three months and < five years and who still experienced difficulties for walking.

Each patient will receive 3 months of intervention targeting their non affected leg. Half of the subjects will have to wear braces with additional weights at the non affected ankle during the day ( > 6 hours), while the other half will wear a similar brace but without weight.

A six minutes walking test will be given before and after the intervention, as well six and twelve months later to measure the effect of these interventions. The investigators hypothesize that people receiving the additional weights to the non paretic leg will show greater improvements in their walk abilities.

ELIGIBILITY:
Inclusion Criteria:

* Hemiparesis following ischemic or hemorrhagic infarct of a single hemisphere
* First episode of stroke experienced > 3 months and < 5 years prior to study enrolment
* Functional Ambulation Categories (FAC) score > 3 < 8
* Be able to walk few meters without physical assistance
* Able to understand and follow instructions

Exclusion Criteria:

* Following inpatient physical rehabilitation
* Experienced more than 2 falls during 3 months prior inclusion
* Signs of bilateral impairments
* Daily use of a wheelchair to move
* Contra-indications for daily walk
* Currently participating in any clinical trial with a experimental walking intervention
* Severe arthrosis
* Dementia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2013-05-17 (Actual); Primary Completion 2016-09-08 (Actual); Study Completion 2016-09-08 (Actual)

PRIMARY OUTCOMES:
Six minutes walking test | 3 months after the inclusion
  Total distance walked in meters (6MWD) within the 6 minutes.

SECONDARY OUTCOMES:
six minutes walking test | 6 months after the inclusion
  Total distance walked in meters (6MWD) within the 6 minutes
six minutes walking test | 12 months after the inclusion
  Total distance walked in meters (6MWD) within the 6 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Philippe Regnaux, PhD, Study Director — French School of Public Health (EHESP)
Locations (1):
- Sainte Anne Hospital, Paris, France